CLINICAL TRIAL: NCT03775460
Title: Methotrexate and Prednisolone Study in Erythema Nodosum Leprosum (MaPS in ENL
Brief Title: Methotrexate and Prednisolone Study in Erythema Nodosum Leprosum
Acronym: MaPs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Dr. Soetomo General Hospital (Other Government); The Leprosy Mission Trust, India (Unknown); Alert Hospital, Ethiopia (Other); The Leprosy Mission Bangladesh (Other); Bombay Leprosy Project, India (Unknown); Oswaldo Cruz Foundation (Other); Leprosy Research Initiative (Unknown); The Leprosy Mission Nepal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15762
Record Dates: First submitted 2018-11-29; First posted 2018-12-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-10

CONDITIONS: Erythema Nodosum Leprosum
Keywords: Erythema Nodosum Leprosum; ENL; corticosteroids; Methotrexate; ENL severity scale; quality of life; Leprosy
MeSH Terms: conditions — Leprosy | interventions — Methotrexate; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Placebo Comparator): Participants will receive placebo+ prednisolone. Participants will start receiving 4 dummy tablets per week, than participants weighing less than 60 kg will receive 6 dummy tablets from week 8. The placebo will be prescribe weekly. Participants weighing 60 kg or more will receive 8 dummy tablets from week 8. Participants will receive dummy tablets for 52 weeks. Along with prednisolone. The start dose of prednisolone will be 40 mg per day decreasing dosage for 20 weeks.
  Interventions: Drug: Placebo; Drug: Prednisolone
- intervention (Experimental): Participants will receive Methotrexate(MTX)+prednisolone. All participants in intervention arm will receive an initial dose of MTX 10 mg. The MTX will be increased to 15 mg the following week. Participants weighing less than 60 kg will continue to receive 15 mg of MTX weekly thereafter. Individuals weighing 60 kg or more will receive MTX 20 mg from week 8. At week 48 the MTX will be reduced to 10 mg for two weeks followed by 5 mg for two weeks and then stopped. In total participants will receive 52 weeks of MTX along side prednisolone, which will be the same as the control arm.
  Interventions: Drug: Methotrexate; Drug: Prednisolone

INTERVENTIONS:
Drug: Methotrexate — Participants in the intervention group will receive methotrexate along side prednisolone
  Arms: intervention
Drug: Placebo — Participants in the control arm will receive placebo along side prednisolone
  Arms: control
Drug: Prednisolone — Participants in both arm will receive prednisolone, which will be the same dosage: 40 mg (initial dose) decreasing dosage for 20 weeks

SUMMARY:
Erythema Nodosum Leprosum (ENL) is a painful, debilitating complication of leprosy. Patients often require high doses of corticosteroids for prolonged periods. Thalidomide is expensive and not available in most countries. The use of corticosteroids for long periods is associated with adverse effects and mortality. It is a priority to identify alternative agents to treat ENL. Methotrexate (MTX) is a cheap, widely used medication which has been reported to be effective in ENL resistant to steroids and thalidomide.

DETAILED DESCRIPTION:
This is a double blind randomized controlled trial (RCT) to test the efficacy of MTX for managing ENL. Patients diagnosed with moderate or severe ENL at ENLIST Group centres in Bangladesh, Brazil, Ethiopia, India, Indonesia and Nepal will be randomly allocated to receive a 15 or 20 mg of oral MTX each week for 48 weeks and prednisolone 40 mg per day reducing to zero over 20 weeks. The control group will receive an identical prednisolone scheme. The participants will be stratified into two groups, those with acute ENL, those with chronic/recurrent ENL. The interventions for both populations are the same, although analysed separately. Adverse effects (AE) will be closely monitored clinically and using laboratory tests. Participants will receive folic acid, 5mg daily for 52 weeks except on the day of MTX to prevent AEs, and nausea will be managed with ondansetron.

ELIGIBILITY:
Inclusion Criteria:: ALL OF THE FOLLOWING SIX CRITERIA MUST BE MET IN ORDER FOR AN INDIVIDUAL TO BE ELIGIBLE (ONLY ONE OF 6A TO 6D NEED BE MET):

1. Individuals who diagnosed with leprosy complicated by ENL
2. Individuals with ENL aged 18-60 years old
3. Individuals with ENL deteriorating symptoms
4. Individuals with 10 or more tender, papular or nodular ENL skin lesions
5. Individuals with an EESS score of at least 9
6. Individuals with ENL on:

   1. No current anti- ENL treatment
   2. Prednisolone up to 30mg per day (if ACUTE) or Prednisolone 10-30mg (inclusive) per day (if RECURRENT/ CHRONIC) or equivalent alternative corticosteroid dose OR
   3. Thalidomide or other non-steroidal anti-ENL medication OR
   4. A combination of prednisolone (up to 30mg) and another non-steroidal anti-ENL medication (thalidomide, clofazimine, azathioprine, pentoxifylline, ciclosporin, minocycline)

Exclusion criteria:

1. Individuals who were first diagnosed with ENL more than 4 years prior to enrolment
2. Individuals less than 18 years old or older than 60 years
3. Individuals weighing less than 35kg
4. Individuals with 9 or fewer tender, popular or nodular ENL skin lesions
5. Individuals with an EESS score of 8 or less
6. Women of child bearing capacity who decline to use two forms of adequate contraception and men who decline to use two forms of adequate contraception
7. Pregnant or breastfeeding women
8. Individuals with recurrent or chronic ENL who deteriorate on a dose of prednisolone less than 10 mg or more than 30 mg
9. Individuals who have taken methotrexate by any route for the last 12 weeks
10. Individuals with a hypersensitivity to methotrexate or a recognised contraindication ( please see Methotrexate information sheet)
11. Individuals currently diagnosed with Type 1 reaction or Lucio's phenomenon
12. Individuals with the severe abnormalities in screening investigations
13. Positive serology for HIV, Hepatitis B or C
14. Evidence of tuberculosis or pulmonary fibrosis
15. A history of chronic liver disease or excessive alcohol or illicit substance consumption
16. Individuals with severe inter-current infections, uncontrolled diabetes, active peptic ulcer disease, untreated malignancy
17. Individuals unable to attend regularly for assessment or monitoring

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals free from Erythema Nodosum Leprosum (ENL) flares in 24 weeks | During the first 24 weeks
  Proportion of individuals who have not required additional prednisolone during the first 24 weeks. The aim is to evaluate if individuals in the methotrexate regimen will need less prednisolone than the control arm.
Proportion of individuals free from ENL flares in 48 weeks | During first 48 weeks
  Proportion of individuals who have not required additional prednisolone during the first 48 weeks. To evaluate if methotrexate will be more efficient to control ENL than only prednisolone

SECONDARY OUTCOMES:
Change in ENLIST ENL severity scale score (EESS) | 60 weeks
  ENLIST group (Erythema Nodosum Leprosum International STudy) developed and validated a severity scale for ENL, which consist 10 symptoms and signs of ENL and range from 0 to 30 points. Mild ENL is categorised as an score of 8 or less. We will measure the change in ENLIST ENL Severity Scale score from baseline to the first flare of ENL requiring additional prednisolone
Quality of life changes: 36- Item Short Form (SF-36) questionnaire | at 24 and 48 weeks
  Change in patient reported health-related quality of life at 24 and 48 weeks from baseline. This will be measured by 36- Item Short Form (SF-36) questionnaire developed by RAND, validated worldwide. The SF-36 consists of 8 scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability. If the score is 0 is equivalent to maximum disability. The 8 sections are vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, emotional role functioning, social role functioning and mental health.
Quality of life changes regarding skin condition: Dermatology life quality Index (DLQI) | at 24 and 48 weeks
  Change in patient reported health-related quality of life at 24 and 48 weeks, specific to skin condition, such as ENL. It will be used the Dermatology life quality Index (DLQI),which is a questionnaire of 10 questions to specific evaluate quality of life in dermatologic conditions.The score can range from 0 to 30, meaning 0 no effect at all on patient's life to 30 extremely large effect on patient's life.
Proportion of individuals free from ENL flares at 60 weeks | 60 weeks
  Proportion of individuals who do not require prednisolone at 60 weeks
ENL flares per individual up to 60 weeks | 60 weeks
  Number of flares of ENL per individual requiring additional prednisolone up to 60 weeks
Severity of ENL flares | 60 weeks
  As stated on outcome 3, the severity of ENL will be measured by ENLIST ENL severity scale. The scale is composed by 10 symptoms and signs of ENL and range from 0 to 30 points. Mild ENL is categorised as an score of 8 or less. We will measure the maximum severity of flares of ENL requiring additional prednisolone up to 60 weeks
Time to the first flare of ENL | 60 weeks
  How long it takes to a participant who has an ENL flare to present with first episode of flare after enrolment
Adverse effects | 60 weeks
  Proportion of individuals with treatment related adverse effects
Quality of life at 60 weeks: SF-36 questionnaire | 60 weeks
  As described on outcome 4. We will use SF-36 questionnaire to measure quality of life. Change in patient reported health-related quality of life at 60 weeks from baseline
Quality of life at 60 weeks regarding skin condition: Dermatology Life Quality Index (DLQI) questionnaires | 60 weeks
  As described on outcome 5. We will use DLQI questionnaires to measure quality of life. Change in patient reported health-related quality of life at 60 weeks from baseline, specific to skin conditions such as ENL.
Individuals free from ENL flares in 60 weeks | 60 weeks
  Proportion of individuals who have not required additional prednisolone in the 60 weeks of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Walker, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (7):
- TMLI Bangladesh/ DBLM hospital, Dhaka, Bangladesh
- FIOCRUZ, Rio de Janeiro, Brazil
- ALERT, Addis Ababa, Ethiopia
- India (2):
  - The Leprosy Mission Trust, Delhi
  - Bombay Leprosy Project, Mumbai
- Soetomo Hospital, Surabaya, Indonesia
- Anandaban Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambert SM, Nigusse SD, Alembo DT, Walker SL, Nicholls PG, Idriss MH, Yamuah LK, Lockwood DN. Comparison of Efficacy and Safety of Ciclosporin to Prednisolone in the Treatment of Erythema Nodosum Leprosum: Two Randomised, Double Blind, Controlled Pilot Studies in Ethiopia. PLoS Negl Trop Dis. 2016 Feb 26;10(2):e0004149. doi: 10.1371/journal.pntd.0004149. eCollection 2016 Feb. PMID 26919207
- [Background] Pocaterra L, Jain S, Reddy R, Muzaffarullah S, Torres O, Suneetha S, Lockwood DN. Clinical course of erythema nodosum leprosum: an 11-year cohort study in Hyderabad, India. Am J Trop Med Hyg. 2006 May;74(5):868-79. PMID 16687695
- [Background] Kumar B, Dogra S, Kaur I. Epidemiological characteristics of leprosy reactions: 15 years experience from north India. Int J Lepr Other Mycobact Dis. 2004 Jun;72(2):125-33. doi: 10.1489/1544-581X(2004)0722.0.CO;2. PMID 15301592
- [Background] Chandler DJ, Hansen KS, Mahato B, Darlong J, John A, Lockwood DN. Household costs of leprosy reactions (ENL) in rural India. PLoS Negl Trop Dis. 2015 Jan 15;9(1):e0003431. doi: 10.1371/journal.pntd.0003431. eCollection 2015 Jan. PMID 25590638
- [Background] Walker SL, Lebas E, Doni SN, Lockwood DN, Lambert SM. The mortality associated with erythema nodosum leprosum in Ethiopia: a retrospective hospital-based study. PLoS Negl Trop Dis. 2014 Mar 13;8(3):e2690. doi: 10.1371/journal.pntd.0002690. eCollection 2014 Mar. PMID 24625394
- [Background] Walker SL, Waters MF, Lockwood DN. The role of thalidomide in the management of erythema nodosum leprosum. Lepr Rev. 2007 Sep;78(3):197-215. PMID 18035771
- [Background] Walker SL, Sales AM, Butlin CR, Shah M, Maghanoy A, Lambert SM, Darlong J, Rozario BJ, Pai VV, Balagon M, Doni SN, Hagge DA, Nery JAC, Neupane KD, Baral S, Sangma BA, Alembo DT, Yetaye AM, Hassan BA, Shelemo MB, Nicholls PG, Lockwood DNJ; Erythema Nodosum Leprosum International STudy Group. A leprosy clinical severity scale for erythema nodosum leprosum: An international, multicentre validation study of the ENLIST ENL Severity Scale. PLoS Negl Trop Dis. 2017 Jul 3;11(7):e0005716. doi: 10.1371/journal.pntd.0005716. eCollection 2017 Jul. PMID 28671966
- [Background] Wemambu SN, Turk JL, Waters MF, Rees RJ. Erythema nodosum leprosum: a clinical manifestation of the arthus phenomenon. Lancet. 1969 Nov 1;2(7627):933-5. doi: 10.1016/s0140-6736(69)90592-3. No abstract available. PMID 4186599
- [Background] Moraes MO, Sarno EN, Almeida AS, Saraiva BC, Nery JA, Martins RC, Sampaio EP. Cytokine mRNA expression in leprosy: a possible role for interferon-gamma and interleukin-12 in reactions (RR and ENL). Scand J Immunol. 1999 Nov;50(5):541-9. doi: 10.1046/j.1365-3083.1999.00622.x. PMID 10564558
- [Background] Kahawita IP, Lockwood DN. Towards understanding the pathology of erythema nodosum leprosum. Trans R Soc Trop Med Hyg. 2008 Apr;102(4):329-37. doi: 10.1016/j.trstmh.2008.01.004. Epub 2008 Mar 3. PMID 18313706
- [Background] Narayanan RB, Laal S, Sharma AK, Bhutani LK, Nath I. Differences in predominant T cell phenotypes and distribution pattern in reactional lesions of tuberculoid and lepromatous leprosy. Clin Exp Immunol. 1984 Mar;55(3):623-8. PMID 6423326
- [Background] Sarno EN, Grau GE, Vieira LM, Nery JA. Serum levels of tumour necrosis factor-alpha and interleukin-1 beta during leprosy reactional states. Clin Exp Immunol. 1991 Apr;84(1):103-8. PMID 2015700
- [Background] Barnes PF, Chatterjee D, Brennan PJ, Rea TH, Modlin RL. Tumor necrosis factor production in patients with leprosy. Infect Immun. 1992 Apr;60(4):1441-6. doi: 10.1128/iai.60.4.1441-1446.1992. PMID 1548069
- [Background] Polycarpou A, Walker SL, Lockwood DN. A Systematic Review of Immunological Studies of Erythema Nodosum Leprosum. Front Immunol. 2017 Mar 13;8:233. doi: 10.3389/fimmu.2017.00233. eCollection 2017. PMID 28348555
- [Background] Hossain D. Using methotrexate to treat patients with ENL unresponsive to steroids and clofazimine: a report on 9 patients. Lepr Rev. 2013 Mar;84(1):105-12. PMID 23741889
- [Background] Kar BR, Babu R. Methotrexate in resistant ENL. Int J Lepr Other Mycobact Dis. 2004 Dec;72(4):480-2. doi: 10.1489/1544-581X(2004)722.0.CO;2. PMID 15755203
- [Background] Rahul N, Sanjay KS, Singh S. Effectiveness of Methotrexate in prednisolone and thalidomide resistant cases of Type 2 lepra reaction: report on three cases. Lepr Rev. 2015 Dec;86(4):379-82. No abstract available. PMID 26964434
- [Background] Sousa AL, Fava VM, Sampaio LH, Martelli CM, Costa MB, Mira MT, Stefani MM. Genetic and immunological evidence implicates interleukin 6 as a susceptibility gene for leprosy type 2 reaction. J Infect Dis. 2012 May 1;205(9):1417-24. doi: 10.1093/infdis/jis208. Epub 2012 Mar 29. PMID 22459738
- [Background] Shannon E, Noveck R, Sandoval F, Kamath B, Kearney M. Thalidomide suppressed interleukin-6 but not tumor necrosis factor-alpha in volunteers with experimental endotoxemia. Transl Res. 2007 Nov;150(5):275-80. doi: 10.1016/j.trsl.2007.05.003. Epub 2007 Jun 26. PMID 17964516
- [Background] Rajappa M, Rathika S, Munisamy M, Chandrashekar L, Thappa DM. Effect of treatment with methotrexate and coal tar on adipokine levels and indices of insulin resistance and sensitivity in patients with psoriasis vulgaris. J Eur Acad Dermatol Venereol. 2015 Jan;29(1):69-76. doi: 10.1111/jdv.12451. Epub 2014 Mar 25. PMID 24665910
- [Background] Martiniuk F, Giovinazzo J, Tan AU, Shahidullah R, Haslett P, Kaplan G, Levis WR. Lessons of leprosy: the emergence of TH17 cytokines during type II reactions (ENL) is teaching us about T-cell plasticity. J Drugs Dermatol. 2012 May;11(5):626-30. PMID 22527432
- [Background] Li Y, Jiang L, Zhang S, Yin L, Ma L, He D, Shen J. Methotrexate attenuates the Th17/IL-17 levels in peripheral blood mononuclear cells from healthy individuals and RA patients. Rheumatol Int. 2012 Aug;32(8):2415-22. doi: 10.1007/s00296-011-1867-1. Epub 2011 Jun 21. PMID 21691744
- [Background] Reinhold-Keller E, de Groot K. Use of methotrexate in ANCA-associated vasculitides. Clin Exp Rheumatol. 2010 Sep-Oct;28(5 Suppl 61):S178-82. Epub 2010 Oct 28. PMID 21044456
- [Background] Marzano AV, Ishak RS, Saibeni S, Crosti C, Meroni PL, Cugno M. Autoinflammatory skin disorders in inflammatory bowel diseases, pyoderma gangrenosum and Sweet's syndrome: a comprehensive review and disease classification criteria. Clin Rev Allergy Immunol. 2013 Oct;45(2):202-10. doi: 10.1007/s12016-012-8351-x. PMID 23334898
- [Background] Davatchi F, Shams H, Shahram F, Nadji A, Chams-Davatchi C, Sadeghi Abdollahi B, Faezi T, Akhlaghi M, Ashofteh F. Methotrexate in ocular manifestations of Behcet's disease: a longitudinal study up to 15 years. Int J Rheum Dis. 2013 Oct;16(5):568-77. doi: 10.1111/1756-185X.12139. Epub 2013 Jul 4. PMID 24164845
- [Background] Warren RB, Griffiths CE. The potential of pharmacogenetics in optimizing the use of methotrexate for psoriasis. Br J Dermatol. 2005 Nov;153(5):869-73. doi: 10.1111/j.1365-2133.2005.06880.x. PMID 16225593
- [Background] Warren RB, Griffiths CE. Systemic therapies for psoriasis: methotrexate, retinoids, and cyclosporine. Clin Dermatol. 2008 Sep-Oct;26(5):438-47. doi: 10.1016/j.clindermatol.2007.11.006. PMID 18755362
- [Background] Dalrymple JM, Stamp LK, O'Donnell JL, Chapman PT, Zhang M, Barclay ML. Pharmacokinetics of oral methotrexate in patients with rheumatoid arthritis. Arthritis Rheum. 2008 Nov;58(11):3299-308. doi: 10.1002/art.24034. PMID 18975321
- [Background] Kaur I, Dogra S, Narang T, De D. Comparative efficacy of thalidomide and prednisolone in the treatment of moderate to severe erythema nodosum leprosum: a randomized study. Australas J Dermatol. 2009 Aug;50(3):181-5. doi: 10.1111/j.1440-0960.2009.00534.x. PMID 19659979
- [Background] Warren RB, Weatherhead SC, Smith CH, Exton LS, Mohd Mustapa MF, Kirby B, Yesudian PD. British Association of Dermatologists' guidelines for the safe and effective prescribing of methotrexate for skin disease 2016. Br J Dermatol. 2016 Jul;175(1):23-44. doi: 10.1111/bjd.14816. No abstract available. PMID 27484275
- [Background] World Health Organization. WHO Expert Committee on Leprosy. World Health Organ Tech Rep Ser. 2012;(968):1-61, 1 p following 61. PMID 22970604
- [Background] Warren RB, Mrowietz U, von Kiedrowski R, Niesmann J, Wilsmann-Theis D, Ghoreschi K, Zschocke I, Falk TM, Blodorn-Schlicht N, Reich K. An intensified dosing schedule of subcutaneous methotrexate in patients with moderate to severe plaque-type psoriasis (METOP): a 52 week, multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Feb 4;389(10068):528-537. doi: 10.1016/S0140-6736(16)32127-4. Epub 2016 Dec 22. PMID 28012564
- [Background] Reich K, Langley RG, Papp KA, Ortonne JP, Unnebrink K, Kaul M, Valdes JM. A 52-week trial comparing briakinumab with methotrexate in patients with psoriasis. N Engl J Med. 2011 Oct 27;365(17):1586-96. doi: 10.1056/NEJMoa1010858. PMID 22029980